CLINICAL TRIAL: NCT06341985
Title: Prospective Multicenter Cohort Study for the Analysis of Correlation Between Dosimetric Parameters and RANV (Radiation Associated Nausea and Vomiting) in Patients With Head and Neck Cancer Undergoing Exclusive Radiotherapy (RT)
Brief Title: DOsimetry and Radiation Induced NAusea in Head and Neck Cancers
Acronym: DORIAN
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1593
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Exclusive Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Exclusive Radiotherapy Treatment: Curative radiotherapy treatment using 3 Dimension (3D) conformal or Intensity Modulated Radiation Therapy (IMRT) techniques.
  Interventions: Radiation: Exclusive radiotherapy

INTERVENTIONS:
Radiation: Exclusive radiotherapy — Curative radiotherapy treatment using 3D conformal or Intensity Modulated Radiation Therapy (IMRT) techniques.

SUMMARY:
This is a prospective cohort study for the analysis of correlation between dosimetric parameters and RANV (Radiation Associated Nausea and Vomiting) in patients with head and neck cancer undergoing exclusive radiotherapy (RT).

The primary purpose of this study is to search for a potential correlation between dosimetry and physician- and patient-rated symptoms in patients treated with exclusive radiotherapy for head and neck cancer.

DETAILED DESCRIPTION:
The use of Intensity Modulated Radiation Therapy (IMRT) has become increasingly common in clinical practice for the treatment of head and neck tumors. Despite the well-documented dosimetric advantages of IMRT, there has been a gradual recognition of toxicity profiles that are characteristic and distinct from those known in the era of 2D and 3D techniques, associated with the so-called "dose bath" typical of all intensity-modulated treatments. Among these, one of the main concerns is Radiation-Associated Nausea and Vomiting (RANV), the persistence and severity of which can significantly compromise the quality of life for patients.

Consequently, there has been a growing need to more thoroughly assess the clinical and dosimetric risk factors associated with the onset of RANV in this population. Although several authors have already investigated this aspect, most studies available to date consider cases where concurrent chemotherapy administration may affect the assessment of the outcomes of interest. Even when exclusively focusing on studies centered on IMRT (without concurrent chemotherapy), the generalization of results is at least partially affected by the fact that these are retrospective series with a relatively small population (23-130 patients).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Diagnosis of primary head and neck neoplasm in the following subsites: oropharynx, nasopharynx, oral cavity, paranasal sinuses, salivary glands, and neoplasms with an unknown primary focus.
* Curative radiotherapeutic treatment with photons or protons using 3D conformal or Intensity Modulated Radiation Therapy (IMRT), Volumetric Modulated Arc Therapy (VMAT), Tomotherapy; both photon and proton treatments are allowed.
* Ability to prospectively collect and anonymously submit clinical data related to the patient, pathology, and treatment characteristics (including the radiotherapy treatment plan in RT.dose format) to a single referring center.
* Ability to prospectively collect and anonymously submit DICOM (Digital Imaging and COmmunication in Medicine) files related to pre-RT magnetic resonance imaging (MRI) to a single referring center.
* Ability to collect acute toxicity data (mucositis, xerostomia, nausea, vomiting, weight loss) during radiotherapy and at three months post-treatment.
* Ability to undergo a clinical follow-up examination three months after the completion of radiotherapy.
* Willingness to provide written informed consent for the anonymous use of data for research purposes.

Exclusion Criteria:

* Patients undergoing chemotherapy treatment (neoadjuvant or concurrent with radiotherapy).
* Patients with local and/or locoregional recurrence of head and neck disease.
* Patients previously treated with oncologic interventions in the head and neck region.
* Patients with synchronous distant metastases at the time of diagnosis.
* Inability to comprehensively collect baseline data related to the patient, pathology, and treatment characteristics (including the treatment plan) and follow-up data.
* Inability to obtain written informed consent for the anonymous use of data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck neoplasms (early or locally advanced stage) treated solely with curative radiotherapy, having undergone contrast-enhanced magnetic resonance imaging (MRI), and for whom acute toxicity data are available.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of nausea (acute toxicity) using CTCAE V5.0 | 3 months
  Dose-response correlation between central nervous system (CNS) structures and substructures and nausea (Nausea will be scored using Common Terminology Criteria for Adverse Events- CTCAE- v 5.0

SECONDARY OUTCOMES:
Evaluation of nausea (acute toxicity) using M.D. Anderson Symptom Inventory (MDASI-SCORE) questionnaire | 3 months
  Dose-response correlation between central nervous system (CNS) structures and substructures and nausea evaluated by MDASI-CORE questionnaire
Identification of the organs at risk most strongly correlated with the onset of nausea | 3 months
  Identification of the organs at risk most strongly correlated with the onset of nausea, both through the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (physician-rated outcome) and the MDASI-CORE questionnaire (patient-reported outcomes)
Identification of dosimetric cutoffs for the onset of nausea | 3 months
  Identification of dosimetric cutoffs for the onset of nausea using Normal Tissue Complication Probability (NTCP) models
Comparison of dosimetric analysis between 3D conformal, IMRT and proton therapy techniques | 3 months
  Dosimetric analysis comparing 3D conformal, IMRT, and proton therapy techniques, with a specific focus on the onset of nausea. Evaluation will be conducted using both the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and the MDASI-CORE questionnaire
Development of machine-learning predictive models for the onset of nausea | 1 year
  Development of machine-learning predictive models for the onset of nausea, incorporating clinical, dosimetric, and imaging parameters

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Volpe, MD, Principal Investigator — European Institute of Oncology
Locations (14):
- Italy (14):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Ospedale "Mons. Dimiccoli", Barletta
  - Azienda Ospedaliera S.Pio, Benevento
  - Ospedale MultiMedica, Castellanza
  - IRCCS Ospedale Policlinico San Martino, Genova
  - European Institute of Oncology, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero-Universitaria di Modena, Modena
  - Azienda Ospedaliero Universitaria Ospedale Maggiore della Carità di Novara, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Complesso Ospedaliero San Giovanni - Addolorata, Roma
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma
  - Ospedale San Giovanni Calibita Fatebenefratelli Isola Tiberina, Roma
  - I.R.C.C.S. MultiMedica - Sesto San Giovanni, Sesto San Giovanni